CLINICAL TRIAL: NCT01601990
Title: A Multicenter, Multinational, Randomized, Placebo-controlled, Parallel Group, Double-blind, Phase 3 Trial to Evaluate the Efficacy and Safety of LC15-0444 in Patients With Type 2 Diabetes
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of LC15-0444 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-DPCL005
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo group(once daily)
- LC15-0444 (Experimental)
  Interventions: Drug: LC15-0444 50mg qd

INTERVENTIONS:
Drug: Placebo group(once daily) — eligible patients were randomized to LC15-0444 50mg or placebo groups and received the assigned treatment for 24 weeks.
  Arms: Placebo
Drug: LC15-0444 50mg qd — eligible patients were randomized to LC15-0444 50mg or placebo groups and received the assigned treatment for 24 weeks
  Arms: LC15-0444

SUMMARY:
Double-blind, randomized, multicenter, multinational (South Korea and India), parallel group study The study was divided into three parts: part 1 was started with an initial 2 weeks of exercise/diet program followed by another 2 weeks of single-blind placebo run-in period; part 2 was a double-blind treatment period during which eligible patients were randomized to LC15-0444 50mg or placebo groups and received the assigned treatment for 24 weeks; part 3 was for those patients who completed part 1 & 2 and consented to receive another 28 weeks of treatment with LC15-0444 50mg. Screening tests were performed on the patients who had given the written informed consent. After 2-week exercise/diet program according to the generally recognized guideline, patients took placebo for another 2 weeks while continuing exercise/diet program. When the 2-week placebo run-in period was completed, eligible patients were assigned either to placebo or 50 mg of LC15-0444 with 1:1 ratio. During the total of 24- week treatment period of part 2 after randomization, each patient visited the investigational site at Week 6, 12, 18, and 24. Completing treatment with placebo or LC15-0444 50mg for 24 weeks after randomization, each patient was asked to provide consent to participate in the part 3 of the study where all the patients were to receive LC15-0444 50mg regardless of the treatment received during the part 2 of the study. During 28-week treatment period of the part 3, each patient visited the investigational site at Week 30, 38, 46, and 52. Total study period from screening was 56 weeks per each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes Mellitus
2. Adults between 18 and 75 of age
3. Patients with HbA1c between 7 % and 11 %
4. Patient who had not received any diabetic medications within 6 weeks from screening
5. Patients who signed on the consent form after informed on the object, method, and risks of the clinical study

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus, gestational diabetes, or secondary diabetes
2. Patients who were taking or needed to take any drugs which may affect the control of blood glucose significantly (ex. glucocorticoids)
3. Patients who had experienced myocardial infarction, unstable angina or prior history of coronary artery bypass surgery within 6 months prior to screening, or patients with arrhythmia requiring treatment
4. Patients with NYHA class II-IV congestive heart failure
5. Patients with history of hepatic cirrhosis
6. Patients with renal failure or whose creatinine clearance was less than 60mL/min
7. Patients with dysfunctional thyroid gland (with abnormal level of TSH)
8. Patients with ALT, AST or CPK exceeding 2.5 times of the upper limit of the normal range
9. Patients with BMI below 20 kg/m2 or exceeding 40 kg/m2
10. Patients with history of asthma or major skin allergy
11. Patients taking thyroid hormone, warfarin, dicoumarin or digoxin.
12. Patients with history of hypersensitivity to metformin or biguanides.
13. Patients who took sodium channel blockers in the last 6 weeks prior to Visit 1.
14. Patients who were treated with insulin or glucagon-like peptide-1 (GLP-1) analogue or who took thiazolidinediones (Glitazone) in the last 6 months prior to Visit 1.
15. Patients with other reasons who the investigator decided not to be eligible for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change of HbAlc | from baseline to Week 24

SECONDARY OUTCOMES:
HbA1c Responder Rate | at Week 24
  HbA1c Responder Rate at Week 24: HbA1c <7 %, <6.5 %

CONTACTS AND LOCATIONS:
Overall Officials: Se Hyun Baek, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- LG Life Sciences, Seoul, South Korea